CLINICAL TRIAL: NCT03115411
Title: Prospective Evaluation of Wing Biliary Stent Patency in Patients With Benign Biliary Obstruction
Brief Title: Prospective Evaluation of Winged Biliary Stent Patency in Patients With Benign Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Associate Professor of Medicine, Division of Gastroenterology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 21604
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Biliary Stricture

STUDY DESIGN:
Intervention Model Description: Patients with benign biliary obstruction who meet all inclusion criteria will be approached to consent for placement of a winged biliary stent for 90 days with appropriate laboratory studies and clinical evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Winged stent (Experimental): Placement of Winged stent for management of biliary obstruction. Stent to be placed for 90 days, with laboratory studies and clinical evaluation during this period to assess for stent potency.
  Interventions: Device: Winged biliary stent (ViaDuct™)

INTERVENTIONS:
Device: Winged biliary stent (ViaDuct™) — Placement of winged biliary stent at ERCP for management of benign biliary stricture.

SUMMARY:
Evaluation of ERCP with placement of a winged plastic biliary stent without a lumen for management of benign biliary strictures.

DETAILED DESCRIPTION:
ERCP with plastic stent placement for resolution of biliary obstruction has been the method of choice for many years. However, stent obstruction is a major limitation of this approach. Studies have shown that the conventional tubular type polyethylene stents (CS) with side holes accumulate significant sludge and their mean patency is approximately 90 days.

Thus patients requiring longer term stenting need to undergo stent exchanges every 2-3 months.

Recently, a stent with a star-shaped cross-section has been developed for biliary applications. This FDA approved biliary Wing stent (WS) (ViaDuct™) is a novel plastic biliary stent that lacks a lumen, and is designed to allow bile to flow on the outside of the stent.

The stent which is star shaped in cross section, channels fluid along its winged perimeter.

It has been proposed that the winged stent design with a lack of central lumen obviates the risk of luminal occlusion and that the risk of occlusion, given the presence of multiple external drainage channels, is smaller. Longer term biliary drainage without the need for stent exchange should therefore be possible with these stents.

The primary aim of this study is to prospectively evaluate the patency rate of the winged stent in up to 90 days for patients with benign biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. All patients age 18 or older referred for ERCP for biliary obstruction from stones or benign strictures that have been confirmed based on clinical, laboratory and imaging findings, with an indication for plastic stent placement.

   One or more biliary stents may be placed during the procedure depending on the indication such as a biliary stricture necessitating multiple stent placements for dilation as the standard of care.
2. Expected patient survival of at least 90 days
3. High likelihood of patient follow-up
4. Patient is able to give a written informed consent
5. Patient is willing and able to comply with the study procedures.

Exclusion Criteria:

1. Patients with cholangitis
2. Patients with bile leak
3. Pregnant patients
4. Patients with any contraindication to endoscopic procedure
5. Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit
6. Patients with malignant biliary strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-09-06 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Winged Biliary Stent: Typical biliary stents have a circular, straw-like lumen. Recently, a stent with a star-shaped cross-section and no central lumen has been developed for biliary applications. This FDA approved biliary Wing stent (WS) (ViaDuct™) is a novel plastic biliary stent that lacks a lumen, and is designed to allow bile to flow on the outside of the stent.
  The stent which is star shaped in cross section, channels fluid along its winged perimeter. It has been proposed that the winged stent design with a lack of central lumen obviates the risk of luminal occlusion and that the risk of occlusion, given the presence of multiple external drainage channels, is smaller. Longer term biliary drainage without the need for stent exchange should therefore be possible with these stents.
  in this arm, we utilize the biliary wing stent in standard clinical settings (biliary obstruction) and assess patency
Period: Overall Study
Arm/Group | Winged Biliary Stent
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Winged Stent: Single arm study (winged biliary stent)
Arm/Group | Winged Stent
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patient reported
  Participants
    American Indian or Alaska Native | 0
    Asian | 6
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 12
    More than one race | 3
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Location of procedure (documented)
  participants
    United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Stent Patency at 90 Days
Description: Evaluation of laboratory studies and clinical status to assess for stent patency/evidence of biliary obstruction
Time Frame: 90 days after placement of stent
Population: Patients with biliary obstruction (non-malignant) who underwent ERCP with placement of winged biliary stent.
Measure: Count of Participants; unit: Participants
Arm/Group | Winged Stent
Number analyzed (Participants) | 23
Participants | 22

ADVERSE EVENTS:
Time Frame: 90 day stent potency was assessed
Description: No difference in definitions.
Arm/Group | Winged Stent
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03115411/Prot_SAP_000.pdf